CLINICAL TRIAL: NCT03649997
Title: A Multi-cohort, Randomized Study in Healthy Subjects to Assess the Pharmacokinetics and Safety of Single and Multiple Ascending Doses of JNJ-61393215 (Suspension), and to Assess the Relative Bioavailability, and the Effect of Food on the Pharmacokinetics, of a New Solid Formulation (Capsules) of JNJ-61393215
Brief Title: A Study of Single and Multiple Ascending Doses of JNJ-61393215 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108492; 2018-001944-80 (EudraCT Number); 61393215EDI1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part 1 (Single Ascending Dose [SAD]): Cohort 1 (Experimental): Participants will receive single oral dose of JNJ-61393215 145 milligram (mg) suspension or matching placebo on day 1, under fasted conditions.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 1 SAD: Cohort 2 (Experimental): Participants will receive single oral dose of JNJ-61393215 225 mg suspension or matching placebo on day 1 under fasted conditions. Dose in this cohort will be determined based on safety and PK data of cohort 1.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 2 Cohort 3: Treatment Sequence CDEF (Experimental): Participants will receive single oral dose of JNJ-61393215 30 mg suspension under fasted condition (Treatment C) in Period 1, then participants will receive single oral dose of JNJ-61393215 30 mg capsule under fasted condition (Treatment D) in Period 2, single oral dose of JNJ-61393215 30 mg capsule with high fat/high-calorie breakfast (Treatment E) in Period 3 followed by single oral dose of JNJ-61393215 30 mg capsule with standardized breakfast (Treatment F) in Period 4, on day 1 of each treatment period. There will be a washout period of at least 7 days between study drug intake in subsequent treatment periods.
  Interventions: Drug: JNJ-61393215
- Part 2 Cohort 3: Treatment Sequence DFCE (Experimental): Participants will receive Treatment D in Period 1, then Treatment F in Period 2, then Treatment C in Period 3 followed by Treatment E in Period 4 on Day 1.
  Interventions: Drug: JNJ-61393215
- Part 2 Cohort 3: Treatment Sequence ECFD (Experimental): Participants will receive Treatment E in Period 1, then Treatment C in Period 2, then Treatment F in Period 3 followed by Treatment D in Period 4 on Day 1.
  Interventions: Drug: JNJ-61393215
- Part 2 Cohort 3: Treatment Sequence FEDC (Experimental): Participants will receive Treatment F in Period 1, then Treatment E in Period 2, then Treatment D in Period 3 followed by Treatment C in Period 4 on Day 1.
  Interventions: Drug: JNJ-61393215
- Part 2 Cohort 4: Treatment Sequence GHIJ (Experimental): Participants will receive single oral dose of JNJ-61393215 suspension under fasted condition (Treatment G) in Period 1, then participants will receive single oral dose of JNJ-61393215 capsule under fasted condition (Treatment H) in Period 2, single oral dose of JNJ-61393215 capsule with high fat/high-calorie breakfast (Treatment I) in Period 3 followed by single oral dose of JNJ-61393215 capsule with standardized breakfast (Treatment J) in Period 4, on day 1 of each treatment period. There will be a washout period of at least 7 days between study drug intake in subsequent treatment periods. Dose in this cohort will be based on the results obtained in Part 1.
  Interventions: Drug: JNJ-61393215
- Part 2 Cohort 4: Treatment Sequence HJGI (Experimental): Participants will receive Treatment H in Period 1, then Treatment J in Period 2, then Treatment D in Period G followed by Treatment I in Period 4 on Day 1.
  Interventions: Drug: JNJ-61393215
- Part 2 Cohort 4: Treatment Sequence IGJH (Experimental): Participants will receive Treatment I in Period 1, then Treatment G in Period 2, then Treatment J in Period 3 followed by Treatment H in Period 4 on Day 1.
  Interventions: Drug: JNJ-61393215
- Part 2 Cohort 4: Treatment Sequence JIHG (Experimental): Participants will receive Treatment J in Period 1, then Treatment I in Period 2, then Treatment H in Period 3 followed by Treatment G in Period 4 on Day 1.
  Interventions: Drug: JNJ-61393215
- Part 3 Cohort 5: Multiple Ascending Dose (Experimental): Participants will receive oral JNJ-61393215 145 mg suspension or matching placebo once daily for 7 days under fasted conditions.
  Interventions: Drug: JNJ-61393215; Drug: Placebo
- Part 3 Cohort 6: Multiple Ascending Dose (Experimental): Participants will receive oral JNJ-61393215 225 mg suspension or matching placebo once daily for 7 days under fasted conditions. Dose may be lowered or increased based on the evaluation of safety and PK of Cohort 5. This dose may be the same as the dose chosen for Cohort 2 (Part 1), or it could be different.
  Interventions: Drug: JNJ-61393215; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-61393215 — Participants will be administered JNJ-61393215 in Part 1, 2 and 3 of study as oral suspension.
Drug: Placebo — Participants will be administered JNJ-61393215-matching placebo in Part 1, 2 and 3 of study as oral suspension.
  Arms: Part 1 (Single Ascending Dose [SAD]): Cohort 1; Part 1 SAD: Cohort 2; Part 3 Cohort 5: Multiple Ascending Dose; Part 3 Cohort 6: Multiple Ascending Dose
Drug: JNJ-61393215 — Participants will be administered JNJ-61393215 in Part 1, 2 and 3 of study as capsule.
  Arms: Part 2 Cohort 3: Treatment Sequence CDEF; Part 2 Cohort 3: Treatment Sequence DFCE; Part 2 Cohort 3: Treatment Sequence ECFD; Part 2 Cohort 3: Treatment Sequence FEDC; Part 2 Cohort 4: Treatment Sequence GHIJ; Part 2 Cohort 4: Treatment Sequence HJGI; Part 2 Cohort 4: Treatment Sequence IGJH; Part 2 Cohort 4: Treatment Sequence JIHG

SUMMARY:
The purpose of this 3 part study are; Part 1: to investigate the pharmacokinetic (PK), safety and tolerability of JNJ-61393215 suspension (ascending dose levels) after single oral dose administration under fasted conditions, Part 2: to evaluate the relative bioavailability of a solid JNJ-61393215 capsule formulation compared to a suspension of JNJ-61393215 under fasted conditions, and the effect of food on the PK of the solid JNJ-61393215 capsule formulation, Part 3: to investigate the PK, safety, and tolerability of JNJ-61393215 suspension (ascending dose levels) after 7 days of once daily dosing in under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential
* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) (including QT interval corrected for heart rate according to Fridericia's formula [QTcF] less-than or equal to [<=] 450 milliseconds (ms) for males and <= 470 ms for females) performed at screening
* Before enrollment, female participants must be of non-childbearing potential, defined as: a) Postmenopausal - A postmenopausal state is defined as no menses for 12 months without an alternative medical cause, as documented by medical records or physician's notes; b) Permanently sterile - Permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy
* Body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (inclusive), and body weight < than 50 kg at screening
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic at screening

Exclusion Criteria:

* Clinically significant abnormal values for hematology, biochemistry, or urinalysis at screening as deemed appropriate by the investigator
* Participants has any liver function test (including alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyltransferase [GGT], alkaline phosphatase [ALP], and bilirubin) at screening more than (>)1.5* upper limit of normal (ULN)
* Participants has estimated glomerular filtration rate (eGFR) according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation < 61 milliliter (mL) / minute /1.73 per square meter (m^2) at screening
* Clinically significant abnormal physical examination, vital signs, or 12 lead ECG at screening as deemed appropriate by the investigator
* Known allergies, hypersensitivity, or intolerance to JNJ-61393215 or its excipients (or lactose)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Observed Analyte Concentration (Cmax) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  Cmax is defined as the maximum observed analyte concentration.
Part 1: Time to Reach Maximum Observed Analyte Concentration (Tmax) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Part 1: Area Under the Analyte Concentration-time Curve from Time Zero to the Time of Last Measurable Concentration (AUC[0-last]) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  AUC(0-last) is defined as the area under the analyte concentration-time curve from time 0 to the time of the last measurable (non-below quantification level [non-BQL]) analyte concentration calculated by linear-linear trapezoidal summation.
Part 1: Area Under the Analyte Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  AUC (0-infinity) is defined as the area under the analyte concentration vs. time curve from time 0 to infinite time, calculated as AUC(0-last) + Clast/lambda(z), where Clast is the last observed measurable (non-BQL) analyte concentration.
Part 1: Apparent Terminal Elimination Rate Constant (lambda[z]) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  lambda(z) is estimated by linear regression using the terminal logarithmic (log)-linear phase of the log transformed concentration vs time data.
Part 1: Apparent Elimination Half-Life (t1/2) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  T1/2 is defined as the apparent terminal elimination half-life and is calculated as 0.693/lambda(z).
Part 1: Apparent Oral Clearance (CL/F) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Part 1: Apparent Volume of Distribution (Vdz/F) of JNJ-61393215 Suspension | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours postdose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired analyte concentration of a drug. Apparent volume of distribution after subcutaneous dose (Vz/F) is influenced by the fraction absorbed.
Part 1: Number of Participants with Adverse Events as a Measure of Safety and Tolerability of JNJ 61393215 Suspension | Up to 7 Weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Part 2: Maximum Observed Analyte Concentration (Cmax) of JNJ-61393215 Capsule | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose
  Cmax is defined as the maximum observed analyte concentration.
Part 2: Area Under the Analyte Concentration-time Curve from Time Zero to the Time of Last Measurable Concentration (AUC[0-last]) of JNJ-61393215 Capsule | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose
  AUC(0-last) is defined as the area under the analyte concentration-time curve from time 0 to the time of the last measurable (non-below quantification level [non-BQL]) analyte concentration calculated by linear-linear trapezoidal summation.
Part 2: Area Under the Analyte Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of JNJ-61393215 Capsule | Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours postdose
  AUC(0-infinity) is defined as the area under the analyte concentration vs. time curve from time 0 to infinite time, calculated as AUC(0-last) + Clast/lambda(z), where Clast is the last observed measurable (non-BQL) analyte concentration.
Part 3: Maximum Observed Analyte Concentration (Cmax) of JNJ-61393215 Suspension | Predose, 20, 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6 and 12 hours postdose on Day 1 and Day 7; 24 and 48 hours postdose on Day 7
  Cmax is defined as the maximum observed analyte concentration.
Part 3: Time to Reach Maximum Observed Analyte Concentration (Tmax) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours postdose on Day 1 and Day 7, 24 and 48 hours postdose on Day 7
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Part 3: Area Under the Analyte Concentration-time Curve from Time 0 to 24 Hours (AUC [0-24]) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours postdose on Day 1 and Day 7, 24 hours postdose on Day 7
  Area under the analyte concentration vs time curve from time 0 to 24 hours, calculated by linear-linear trapezoidal summation.
Part 3: Maximum Trough Concentration (Ctrough) of JNJ-61393215 Suspension | Predose on day 1, 2, 3, 4, 5, 6, 7 and 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 24 and 48 hours postdose on Day 7
  Ctrough is defined as the observed analyte concentration just prior to the beginning or at the end of a dosing interval. Ctrough estimation does not include the concentration that occurs just prior to the first dose.
Part 3: Minimum Observed Analyte Concentration (Cmin) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 24 and 48 hours postdose on Day 7
  Cmin is defined as the minimum observed analyte concentration during the dosing interval.
Part 3: Average Analyte Concentration (Cavg) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 12, 24 and 48 hours postdose on Day 7
  Cavg is defined as the value of the average analyte concentration at steady state over the dosing interval.
Part 3: Fluctuation Index (FI) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours postdose on Day 7
  FI is estimated as the percentage fluctuation (variation) between the maximum and minimum analyte concentration at steady state.
Part 3: Volume of Distribution at Steady-State (Vss) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours postdose on Day 7
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time.
Part 3: Apparent Oral Clearance (CL/F) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours postdose on Day 7
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Part 3: Apparent Terminal Elimination Rate Constant (lambda[z]) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours postdose on Day 7
  lambda(z) is estimated by linear regression using the terminal logarithmic (log)-linear phase of the log transformed concentration vs time data.
Part 3: Apparent Elimination Half-Life (t1/2) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours postdose on Day 7
  T1/2 is defined as the apparent terminal elimination half-life and is calculated as 0.693/lambda(z).
Part 3: Peak by Trough Ratio of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours postdose on Day 7
  Peak by trough ratio is defined as the ratio of the maximum observed analyte concentration to the minimum observed analyte concentration.
Part 3: Observed Accumulation Index Based on AUC (AR AUC) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose on Day 1 and 7
  AR AUC is determined after multiple-dose administration and calculated as AUC (0-24h) on day 7 divided by AUC (0-24h) on day 1.
Part 3: Observed Accumulation Index Based on Cmax (ARCmax) of JNJ-61393215 Suspension | Predose, 20 and 40 minutes, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose on Day 1 and 7
  ARCmax is determined after multiple-dose administration and calculated as Cmax on day 7 divided by Cmax on day 1.

SECONDARY OUTCOMES:
Part 2: Number of Participants with Adverse Events as a Measure of Safety and Tolerability of JNJ 61393215 | Up to 8 Weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Groningen, Netherlands